CLINICAL TRIAL: NCT02643433
Title: Immunogenicity of Co-administration of Measles Containing Vaccine and Japanese Encephalitis Alive Vaccines
Brief Title: Immunogenicity of Co-administration of Measles and Japanese Encephalitis Vaccines
Acronym: MR+JE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention, China (Other Government)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Zhejiang Provincial Center for Disease Control and Prevention (Other Government); Hubei Provincial Center for Disease Control and Prevention (Other)
Responsible Party: Principal Investigator, Huaqing Wang, Deputy Director, National Immunization Program, China CDC, Centers for Disease Control and Prevention, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201518
Record Dates: First submitted 2015-12-23; First posted 2015-12-31 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Measles; Rubella; Japanese Encephalitis
Keywords: Immunogenicity; Coadministration; Measles; Rubella; Japanese encephalitis; Vaccine
MeSH Terms: conditions — Measles; Rubella; Encephalitis, Japanese

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MR and JE coadministration group (Experimental): Infants aged 8 months are vaccinated measles-rubella combined vaccine (MR) and Japanese Encephalitis alive vaccine (JE) in different sites at same time.
  Interventions: Biological: Measles-Rubella combined vaccine(MR); Biological: Japanese Encephalitis alive vaccine(JE)
- MR administration alone group (Active Comparator): Infants aged 8 months are vaccinated measles-rubella combined vaccine alone
  Interventions: Biological: Measles-Rubella combined vaccine(MR)

INTERVENTIONS:
Biological: Measles-Rubella combined vaccine(MR) — 0.5ml for each dose,be administered by single use syringe subcutaneously in the lower part of the deltoid area of lateral arm.
Biological: Japanese Encephalitis alive vaccine(JE) — 0.5ml for each dose be administered by single use syringe subcutaneously in the lower part of the deltoid area of lateral arm.
  Arms: MR and JE coadministration group

SUMMARY:
Japanese encephalitis (JE) is the leading cause of viral neurological disease and disability in Asia. A live attenuated vaccine (LJEV) manufactured in China has several advantages over other JE vaccines such as one dose schedule, using for infants, and the cheaper cost. Because the LJEV has been prequalified by the World Health Organization (WHO) in 2013, it will likely be used in other countries, and possibly co-administered with the first dose of measles-containing vaccine (MCV) to ensure early protection and reduce additional vaccination visits.

The evidence for immunogenicity and safety of co-administration of LJEV with MCV is limited. Only one study conducted in the Philippines examining the co-administration of MCV with LJEV among 9 months infants, the results showed the proportion of achieved sero-protection against measles following MCV (96%) was slightly lower than in the MCV-only group (100%), and the measles antibody titres were also slightly lower in the co-administration group. Due to limited evidence available, the WHO position paper of measles vaccines has encouraged further investigation on the possible impact of co-administration of LJEV on measles vaccine effectiveness.

In China, Measles-Rubella combined vaccine (MR) and LJEV is given at 8 months of age nationally. Considering China is reaching towards the goal of measles elimination, it will be important to conduct a study to compare the immunogenicity of MR administered alone or with LJEV, and also evaluate the safety and tolerability of LJEV administered with MR among 8 months infants.

This study is a prospective, randomized, open-label, multi-center study enrolling infants aged 8 months. Basic demographic information of the infant will be taken and blood samples will be collected at enrollment (baseline) and at 6weeks following administration of MR, the measles antibodies will be measured, and compare seroconversion rates to assess for non-inferiority. All infants will be monitored for adverse events after MR.

DETAILED DESCRIPTION:
Primary Objective:

- To determine whether sero-conversion rates against measles after co-administering measles-rubella (MR) vaccine and live attenuated JE vaccine at 8 months old are not lower than sero-conversion rates among those vaccinated with MR vaccine alone.

Secondary Objective:

* Sero-conversion rates against rubella after co-administering of MR vaccine and live attenuated JE vaccine at 8 months old are no less than those vaccinated with MR vaccine alone.
* To describe the incidence of adverse reactions in concurrent group and non-concurrent vaccination group after initial vaccination and during the follow-up period.

Subjects:

- This study will enroll healthy infants who are between 8 months old and 8 months plus two weeks of age.

Study Arms:

* The subjects are divided into two groups: a MR+JE vaccine co-administration group and a MR vaccine only group.
* After obtaining informed consent from parents or legal guardians, the infants will be randomly assigned to one of the two groups mentioned above. Children and family basic demographic information will be collected at enrollment. One blood sample will be taken before vaccination to measure baseline antibody levels and another blood sample 6 weeks (42-48 days) after vaccination to test for measles and rubella antibody response. JE vaccine will be given the MR vaccine only group after the second blood draw. Adverse reactions will be monitored and recorded after MR vaccination and during the follow-up period.

Sampling size:

* Assuming a seropositivity rate of 93% for measles with minimal interference with JE coadministration, and power of 0.90 with a 0.05 significance level (one-tailed), for a non-inferiority margin of 5%, the sample size per group would be 447 and 526 with 15% attrition.
* The total sample size would be around 1052.

Subject Assignment:

* The subjects will be randomly assigned to MR+JE group and MR only group. In order to randomize the two groups among different vaccination clinics, every 8 subjects are allocated to one randomized unit; random code is allocated to MR+JE group and MR only group according to the ratio of 1:1. The subject number in each vaccination clinic is an integer multiple of 8. This arrangement needs to code 132 randomized units, resulting in a total of 1056 subjects, slightly higher than the calculated sample size.
* The 1056 subjects will be allocated to the 2 provinces equally, with 528 subjects in each province. In each province there will be 264 infants in MR+JE group and 264 infants in MR only group.

Standard Operating Procedures in the field:

The specific procedures that the vaccination clinic participating in the project will do to the subjects are as follows:

1. Make a list of the target children in the vaccination clinic, arrange for appointment for vaccination to children of 8 months old.
2. The children's guardians take children to get the vaccination according to the appointment.
3. Recruit the research subject, and sign the informed consent.
4. Fill in "subject screening form", and screen the eligible subject.
5. The first blood sample collection.
6. Assign into the group according to the coding envelope.
7. Corresponding vaccination of MR+JE or MR only according to the grouping information.
8. Observation for 30 minutes after vaccination in the vaccination clinic.
9. Fill in the questionnaire during observation
10. Distribute the "diary card", notify returning it to the vaccination clinic six weeks later.
11. Follow up the health condition and adverse events after vaccination.
12. When the subjects come back to the vaccination clinic 6 weeks later, take the "diary card" back, and check the information.
13. A second blood sample collection.
14. JE vaccine inoculation for MR only group. Observation for 30 minutes.
15. Inform the subjects that this survey is all over.

Statistical Analysis Plan

* Primary statistical analysis will be to compare sero-conversion rates against measles and rubella between MR+JE group and MR only group using non-inferiority criteria.
* Secondary analyses will be to compare measles and rubella antibody titer levels between MR+JE group and MR only group, and to describe adverse reactions in both groups up to 6 weeks after MR vaccination.

Quality Assurance Plan

1. Training Investigators: Administrative and technical personnel at all levels in study areas are required to participate in training on the study objectives, enrollment procedures, data collection, data entry and management, quality control measures, sample handling and transport, and all other operations involved.
2. Supervision and Monitoring: Chinese Center for Disease Control and Prevention (China CDC) will supervise and monitor each province at least two times during the implementation period;, the province (prefecture) will supervise and monitor each county at least two times during implementation period, and the county level will supervise and monitor each vaccination clinic on selected appointment days. The focus of supervision and monitoring will be to observe whether the vaccination clinics strictly follow protocols and procedures and any problems found can be quickly resolved with timely feedback. Any serious and consistent problems will be reported to the higher level, so that corrections can be made at all levels and in all project areas.
3. Sample Management: Samples collected will be stored in secured, locked laboratories, with cold chain equipment, temperature monitoring and recording. The serum samples in tube A and tube B will be separately packaged and transported from county to province, and then to the designated laboratory, to avoid any loss or unexpected accidents.
4. Vaccine Management: This study will use the same vaccines as the vaccines used in the national immunization program. Vaccination clinics will record vaccine types, the number of vaccine doses, and batch number. Expiration dates will be monitored and expired vaccines will not be used.
5. Logistics Support: China CDC will provide sample coding bar, consent form, investigation questionnaire, data collection forms, and operation manual. Provincial / prefecture CDCs will be responsible for provision or procurement of equipment/materials used for blood collection, serum separation, transportation and storage, and laboratory supplies, and to ensure that all materials meet study requirements.

ELIGIBILITY:
Inclusion Criteria:

1. Infants between 8 months and 8 months plus two weeks of age;
2. Complete vaccination of national immunization schedule before 8 months;
3. Healthy infants;
4. Live in the study county with good compliance who can participate in the entire observation period.

Exclusion Criteria:

1. Previous history of measles, rubella, or JE;
2. Previously received vaccines containing measles/rubella or JE components;
3. Contraindications to the study vaccines;
4. Received blood products or immunosuppressive treatments within last 3 months;
5. Received any live attenuated vaccines within the last 4 weeks, or any inactivated vaccines within 2 weeks;
6. Guardian refuses to participate in the study.

Ages: 8 Months to 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1043 (Actual)
Dates: Start 2015-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Seroconversion rate for measles | 6 weeks after vaccination (day 42-48)
  Compare the seroconversion rate of measles antibody between the two groups

SECONDARY OUTCOMES:
Seroconversion rate for rubella | 6 weeks after vaccination (day 42-48)
  Compare the seroconversion rate of rubella antibody between the two groups
Adverse Events Following Immunization | Within 6 weeks after vaccination
  Compare the rate of Adverse Events Following Immunization between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Huaqing Wang, MD, PhD, Principal Investigator — Centers for Disease Control and Prevention, China; Zhijie AN, MD, MPH, Study Director — Centers for Disease Control and Prevention, China; Zijian Feng, MD, MPH, Study Chair — Centers for Disease Control and Prevention, China
Locations (2):
- China (2):
  - Hebei Provincial Center for Disease Control and Prevention, Shijiazhuang, Hebei
  - Zhejiang Provincial Center for Disease Control and Prevention, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
we will share the serum results with the participants after completing laboratory test. and we will publish articles to share our research.

REFERENCES:
- [Background] Gatchalian S, Yao Y, Zhou B, Zhang L, Yoksan S, Kelly K, Neuzil KM, Yaich M, Jacobson J. Comparison of the immunogenicity and safety of measles vaccine administered alone or with live, attenuated Japanese encephalitis SA 14-14-2 vaccine in Philippine infants. Vaccine. 2008 Apr 24;26(18):2234-41. doi: 10.1016/j.vaccine.2008.02.042. Epub 2008 Mar 18. PMID 18394765
- [Background] Measles vaccines: WHO position paper. Wkly Epidemiol Rec. 2009 Aug 28;84(35):349-60. No abstract available. English, French. PMID 19714924
- [Derived] Li Y, Chu SY, Yue C, Wannemuehler K, Xie S, Zhang F, Wang Y, Zhang Y, Ma R, Li Y, Zuo Z, Rodewald L, Xiao Q, Feng Z, Wang H, An Z. Immunogenicity and safety of measles-rubella vaccine co-administered with attenuated Japanese encephalitis SA 14-14-2 vaccine in infants aged 8 months in China: a non-inferiority randomised controlled trial. Lancet Infect Dis. 2019 Apr;19(4):402-409. doi: 10.1016/S1473-3099(18)30650-9. Epub 2019 Mar 1. PMID 30833160